CLINICAL TRIAL: NCT04313075
Title: A Compassionate Use Study of Leronlimab (PRO 140) Plus Treatment of Physician's Choice in Patients With CCR5+ Metastatic Triple Negative Breast Cancer (mTNBC)
Brief Title: A Compassionate Use Study of Leronlimab in Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CD07_TNBC_CompassionateUse
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — leronlimab

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Leronlimab — Leronlimab is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: (PRO 140)

SUMMARY:
This is a single arm, compassionate use study with 30 patients for leronlimab (PRO 140) combined with a treatment of physician's choice (TPC) in patients with CCR5+ mTNBC.

DETAILED DESCRIPTION:
This is a single arm, compassionate use study with 30 patients for leronlimab (PRO 140) combined with a treatment of physician's choice (TPC) in patients with chemokine receptor 5 (CCR5+) mTNBC.

Leronlimab (PRO 140) will be administered subcutaneously as a weekly dose of 350 or 525 mg until disease progression or intolerable toxicity. Treatment of Physician's Choice (TPC) is defined as one of the following single-agent chemotherapy drugs administrated according to local practice: eribulin, gemcitabine, capecitabine, paclitaxel, nab-paclitaxel, vinorelbine, ixabepilone, or carboplatin. The selected treatment should be administered as per the dosing schedule included on the package insert.

In this study, patients will be evaluated for tumor response approximately every 3 months or according to institution's standard practice by computed tomography (CT), positron emission computed tomography (PET/CT) or MRI with contrast (per treating investigator's discretion) using the same method as at baseline. Tumor measurements will be done using RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologically confirmed diagnosis of TNBC. Must demonstrate HER-2 negative (IHC 0, 1+, or fluorescence in situ hybridization (FISH) negative and ER< 1%, and PR < 1%, per ASCO/CAP criteria); Note: Patients with ER and/or PR<10% who have failed on endocrine therapy will also be eligible for participation in the study.
2. Demonstrate CCR5 + by IHC (>10% of primary or metastatic tumor cells shows membranous staining and/or high predominance of CCR5+ tumor-infiltrating leukocytes completed at the reference laboratory of Dr. Hallgeir Rui at medical College of Wisconsin).

   Note: This test will be done as part of the pre-screening period. It will be performed in archival metastatic tissue. If archival tissue is not available then, fresh biopsy will be done;
3. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion (in case archival tissue is not available);
4. Patients with de novo (metastatic or stage IV at initial diagnosis) breast cancer OR Patients with locally recurrent or metastatic breast cancer who have been treated with up to 3 previous line of systemic therapies (including neo/adjuvant setting) and progressed or were intolerant to the latest treatment.

   Note: Patients with programmed cell death ligand-1 (PDL-1+) that elect not to receive checkpoint inhibitor or are excluded for medical conditions will be eligible for participation in the study.
5. Patients must have measurable disease based on RECIST v1.1;
6. Female patients, ≥ 18 years of age;
7. Patients must exhibit a/an ECOG performance status of 0-1;
8. Life expectancy of at least 6 months;
9. Patients must have adequate organ and bone marrow function within 28 days prior to registration, as defined below:

   * leukocytes ≥ 3,000/mcL;
   * absolute neutrophil count ≥ 1,500/mcL;
   * platelets ≥ 100,000/mcL;
   * total bilirubin: within normal institutional limits;
   * AST(SGOT) &ALT(SPGT) ≤ 2.5 X institutional upper limit of normal (ULN) (applicable to all patients, irrespective of liver disease or metastasis); and
   * creatinine: within normal institutional limits.
10. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
11. Females of child-bearing potential (FOCBP) and males must agree to use two medically accepted methods of contraception with hormonal or barrier method of birth control, or abstinence, prior to study entry, for the duration of study participation and for 60 days after the last dose of study drug (Refer to Appendix 1). Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Note: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; and
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months).
12. FOCBP must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
13. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

1. HER-2 overexpressed/amplified Metastatic Breast Cancer (MBC) (Appendix 2 for guidelines from ASCO);
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days prior to enrollment;
3. Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible;
4. Patients who have had prior exposure to CCR5 antagonists are not eligible;
5. Patients who have a known additional malignancy that is progressing or requires active treatment are not eligible. Patients who have had a prior diagnosis of cancer and if it has been <3 years since their last treatment are not eligible. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer;
6. Has an active infection requiring systemic therapy. Note: Patients must complete any treatment with antibiotics prior to registration;
7. Patients who have a known HIV positive status or known/ active Hepatitis B and/or C infection are not eligible;
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note:

   Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial; and
11. Is pregnant or breastfeeding, or expecting to conceive or have children within the projected duration of the trial, starting with the pre-screening or screening visit through the duration of study participation.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender eligibility will be based on self-representation of gender identity.

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT04313075/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04313075/SAP_001.pdf